CLINICAL TRIAL: NCT06436547
Title: The Efficacy and Safety of Subiculum Electrical Stimulation for Temporal Lobe Epilepsy With Bilateral Hippocampal Sclerosis: A Prospective, Single-Arm Pilot Trial
Brief Title: Subiculum Electrical Stimulation for Temporal Lobe Epilepsy With Biliteral Hippocampus Sclerosis(SESTB)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-112-002
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Deep Brain Stimulation; Drug Resistant Epilepsy; Subiculum; Temporal lobe epilepsy with bilateral hippocampal sclerosis; neuromodulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bilateral subiculum-DBS group (Experimental): participants will undergo bilateral subiculum-DBS ON with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.
  Interventions: Device: Subiculum-DBS ON

INTERVENTIONS:
Device: Subiculum-DBS ON — The surgical intervention named deep brain stimulation is a well-established neurosurgical treatment for drug-resistant epilepsy.The targets used in this study are biliteral subiculum.The devices used for intervention have been approved by Chinese National Medical Products Administration (CFDA). The postoperative drug dosage adjustment depends on the efficacy of DBS and the judgment of the epilepsy specialist.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of deep brain stimulation (DBS) of Subiculum as adjunctive therapy for reducing the frequency of seizures in drug-resistant temporal lobe epilepsy with bilateral hippocampal sclerosis

DETAILED DESCRIPTION:
This project aims to include 6 participants, and evaluate the effectiveness and safety of bilateral hippocampal subcortical stimulation in patients with temporal lobe epilepsy and bilateral hippocampal sclerosis through A prospective, interventional, unblinded, single-arm clinical trial. It is expected to provide new therapeutic options for patients with temporal lobe epilepsy and bilateral hippocampal sclerosis with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 14 -65 years of age
* Refractory to anti-seizure medications (ASMs).
* Persistence of disabling seizures at least 3 times per 3 months or greater, and once or more in recent 1 month.
* After comprehensive preoperative evaluation, patients who are considered unsuitable for or refuse resection surgery, or those for whom the effects of epileptic focus resection and thermocoagulation surgery are not satisfactory.
* Participants must have had a non-invasive video-EEG monitoring revealing seizure semiology and ictal EEG consistent with bilateral Temporal Lobe Epilepsy
* Biliteral hippocampal atrophy on MRI T1 imaging with increased ipsilateral mesial signal on T2 imaging
* Informed consent signed.

Exclusion Criteria:

* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations;
* Psychogenic non-epileptic seizures within 12 months;
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., pacemaker, spinal cord stimulator, responsive neurostimulation) or any metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagal nerve stimulators are allowed if the parameter remains stable for at least 3 months prior to the screening visit;
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. (e.g., coagulation abnormalities, etc.) or the need for chronic anticoagulation or antiplatelet aggregation medications;
* IQ < 55 or severe cognitive dysfunction, unable to complete the study;
* Diagnosed with a progressive neurological disorder (including progressive Rasmussen's encephalitis, etc.);
* Diagnosed with a severe neuropsychiatric disorder such as dementia, major depression (admission to a psychiatric specialty/hospital within 5 years or any suicidal or self-injurious tendencies), schizophrenia, or neurodegenerative disorders;
* Diagnosed with other serious physical disorders, internal diseases or severe abnormalities in liver or kidney function;
* Pregnant, or planning to pregnant within 2 years;
* Participation in another clinical study within 3 months;
* Not suitable for enrollment as assessed by the multidisciplinary team of the center.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency (SF28) | Up to 1 year after subculum-DBS
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3-month SF28 in the baseline period. The seizure frequency in open-label phase is defined as SF28 per month during the open-label period. Percent change in seizure frequency=100*(open-label SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 1 year after subculum-DBS
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 1 year after subculum-DBS
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Cognitive function evaluation (MMSE) | Up to 1 year after subculum-DBS
  Percentage change from baseline in Mini-Mental State Examination (MMSE) score.
Cognitive function evaluation (MoCA) | Up to 1 year after subculum-DBS
  Percentage change from baseline in Montreal Cognitive Assessment (MoCA) score.
Adverse Events | Up to 1 year after subculum-DBS
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 1 year after subculum-DBS
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No